CLINICAL TRIAL: NCT06724796
Title: Yoga 4 Body Image (Y4BI): Investigating the Impact of Yoga on Body Image and Eating Behaviours in Young Women
Brief Title: Yoga 4 Body Image (Y4BI): Investigating the Impact of Yoga on Body Image and Eating Behaviours
Acronym: Y4BI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Silvia Cerea, Ph.D., University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 389
Record Dates: First submitted 2024-11-16; First posted 2024-12-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Body Dissatisfaction; Body Image; Eating Behaviors
MeSH Terms: conditions — Feeding Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Y4BI (Experimental): The yoga classes will be conducted once a week, in groups, with each session lasting 1 hour. They will be led by a qualified instructor with over 10 years of teaching experience in yoga.
  Interventions: Other: Y4BI
- ACTIVE (Active Comparator): The total body classes will take place once a week, with each session lasting one hour. They will be led by a kinesiology specialist in preventive and adapted physical activities.
  Interventions: Other: ACTIVE

INTERVENTIONS:
Other: Y4BI — The yoga classes will follow the Iyengar method, one of the most widely practiced traditional yoga styles, aimed at promoting body alignment and precision in executing poses (asanas) through the use of props such as blankets, straps, cushions, chairs, and blocks, making the poses accessible to all individuals.
  The classes will be conducted once a week, in groups, with each session lasting 1 hour. They will be led by a qualified instructor with over 10 years of teaching experience in yoga. The classes will be adapted for beginners who do not practice yoga regularly.
  Arms: Y4BI
Other: ACTIVE — The total body classes will take place once a week, with each session lasting one hour. They will be led by a kinesiology specialist in preventive and adapted physical activities.
  Arms: ACTIVE

SUMMARY:
The practice of yoga can positively impact body image, a psychological construct encompassing perceptual, emotional, cognitive, and behavioral aspects, which can be either positive or negative. Negative body image manifests as extreme dissatisfaction with one's body-a condition particularly common among young women-that places them at significant risk for developing Body Image Disorders (BIDs). In contrast, positive body image is characterized by an overall respect for one's body.

Current research on the impact of yoga on body image has several limitations, making it challenging to determine whether yoga practice truly has a positive effect on body image and to identify the mechanisms underlying this impact. To address these gaps, the present project aims to overcome the limitations of existing studies by investigating the impact of yoga on body image through quantitative methodologies and by exploring the mechanisms that drive this effect.

The project consists of two phases:

1. Investigating the impact of yoga on body image (both positive and negative) and eating behaviours in a population characterized by high levels of body dissatisfaction-young women.
2. Examining the psychological mechanisms underlying yoga's impact on body image, including increased interoceptive awareness, embodiment, and self-compassion, as well as a reduction in self-objectification.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18-35 years old

Exclusion Criteria:

* Regular yoga practice
* Pregnancy
* Medical conditions that preclude yoga practice (e.g., neurodegenerative diseases, recent injuries, rheumatic conditions)
* Full-blown body image disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Negative Body Image | 10 weeks
  Assessed with the Questionario sul Dismorfmismo Corporo (QDC; Cerea et al., 2017), a self-report questionnaire assessing negative body image made up of 40 items.
Body Appreciation | 10 weeks
  Assessed with the Body Appreciation Scale-2 (BAS-2; Tylka & Wood-Barcalow, 2015b, Casale et al., 2021), a self-report questionnaire assessing body appreciation made up of 10 items.
Functionality Appreciation | 10 weeks
  Assessed with the Functionality Appreciation Scale (FAS; Alleva, Tylka & Van Diest, 2017, Cerea et al., 2021), a self-report questionnaire assessing functionality appreciation made up of 7 items.
Dysfunctional Eating Behaviours and Risk of Developing Eating Disorders | 10 weeks
  Assessed with the Eating Disorder Risk Composite Score of the Eating Disorder Inventory-3 (EDI-3; Garner, 2004; Giannini, Pannocchia, Dalla Grave, Muratori & Viglione, 2008), a self-report questionnaire assessing the risk of developing eating disorders
Functional Eating Behaviors | 10 weeks
  Assessed with the Intuitive Eating Scale-2 (IES-2; Tylka & Kroon Van Diest, 2013, Swami et al., 2021), a self-report questionnaire assessing the ability to eat intuitively.

SECONDARY OUTCOMES:
Embodiment | 10 weeks
  Assessed with the Experience of Embodiment Scale (EES; Piran, Teall, & Counsell, 2020), a self-report questionnaire investigating embodiment.
Interoceptive Awareness | 10 weeks
  Assessed with the Multidimensional Assessment of Interoceptive Awareness (MAIA; Mehling et al., 2012; Calì et al., 2015), a self-report questionnaire investigating interoceptive awareness
Self-compassion | 10 weeks
  Assessed with the Self-Compassion Scale (SCS, Neff, 2003; Veneziani et al. 2017), a self-report questionnaire investigating self-compassion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Psychology, University of Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No